CLINICAL TRIAL: NCT03158493
Title: Assessment of qSOFA in the Latin America Sepsis Institute Database
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Collaborators: Latin America Sepsis Institute (Unknown)
Responsible Party: Principal Investigator, Flavia Ribeiro Machado, Professor, Federal University of São Paulo
Other Study IDs: 00691812.3.0000.5505
Record Dates: First submitted 2017-05-15; First posted 2017-05-18 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Recently, the Society of Critical Care Medicine (SCCM) and the European Society of Intensive Care Medicine (ESICM) have published new definitions of sepsis, known as Sepsis 3, based on a fairly robust analysis of large, essentially American, databases. In addition to the new definition, a new screening score was suggested, named quickSOFA (qSOFA). This score is positive if two of three variables are present: respiratory rate higher than 22 ipm, reduced level of consciousness and systolic blood pressure lower than 100 mmHg. Although the receiver operator characteristics (ROC) curves suggest an adequate predictive validity for the new score, a lot of controversy around its sensitivity as a screening tool mainly in settings with high mortality rates. Current national Brazilian data show that sepsis mortality in our country, especially in public hospitals from the Unified Health System (SUS), is very high and well above world mortality. The impact of using the qSOFA in these settings is not known. In this context, the present study aims to evaluate the potential impact of using qSOFA as a screening tool in Brazilian private and public institutions. The hypothesis is that the use of qSOFA as a screening tool will have a low sensitivity. As a consequence, patients with the diagnosis of sepsis, with organ dysfunction, will not be detected by this tool. The hypothesis was also that those patients with a qSOFA negative will have a high mortality rate, mainly in Brazilian public hospitals.

DETAILED DESCRIPTION:
All hospitals in the Latin America Sepsis Institute network were invited to participate. This is a national based quality improvement initiative aiming to improve compliance with the sepsis bundles and mortality. The hospitals were instructed to include all patients that presented with the diagnosis of sepsis or septic shock in the emergency department (ED), wards or ICU. The diagnosis of sepsis was based on the previous criteria used by the network, which means presence of suspected infection and an infection-associated organ dysfunction. Organ dysfunction was defined by the presence of any of the following: systolic blood pressure <90 mmHg or mean arterial pressure <65 mmHg or fall in systolic blood pressure> 40 mmHg; creatinine> 2.0 mg / dl or diuresis less than 0.5 ml/kg/h in the last 2 hours, bilirubin> 2mg/dl, platelet count<100,000, lactate> 2 mmol/dl (or above the reference value), coagulopathy (RNI> 1.5 or APTT>60 sec), PaO2/FiO2 ratio <300 or recent or increased O2 need to maintain SpO2> 90. Suspected of infection was based on the clinical suspicious by the attending physician. All patients under end-of-life care and those previously included in the database in the same hospital admission were excluded.

The case managers were instructed to collect the 3 components of the qSOFA criteria, namely reduced level of consciousness, respiratory rate higher than 22 bpm and systolic blood pressure lower than 100 mmHg). In patients included from the ED, these components were checked at the time of triage. In patients in the wards or in the ICU, the 3 components were considered if presented any time in the 24 hours prior to the diagnosis of sepsis.

Outcomes Primary outcome was hospital mortality. Secondary endpoints included admission to ICU and length of ICU stay of more than 48 hours. A secondary composite outcome was hospital mortality plus ICU length of stay higher than two days (for those admitted to the ICU).

ELIGIBILITY:
Inclusion Criteria:

* Suspected source of infection
* Presence of any of the following organ dysfunction

  * Systolic blood pressure <90 mmHg or mean arterial pressure <65 mmHg or fall in systolic blood pressure> 40 mmHg.
  * Creatinine> 2.0 mg / dl or diuresis less than 0.5 ml/kg/h in the last 2 hours OR
  * Bilirubin> 2mg/dl,
  * Platelet count<100,000,
  * Lactate> 2 mmol/dl (or above the reference value),
  * Coagulopathy (RNI> 1.5 or APTT>60 sec),
  * PaO2/FiO2 ratio <300 or recent or increased O2 need to maintain SpO2> 90

Exclusion Criteria:

* End of life care
* Previous sepsis episode in the same hospital admission

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with sepsis and sepsis shock, defined by the presence of any organ dyfunctionn
Sampling Method: Probability Sample
Enrollment: 8435 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Hospital mortality | From date of inclusion through study completion, assessed up to 100 months
  mortality at hospital

SECONDARY OUTCOMES:
admission to ICU in the first 24 hours of the diagnosis of sepsis | From date of inclusion until 24 hours after the diagnosis of sepsis, assessed up to 24 hours after the diagnosis of sepsis
  number of patients who were admitted in the intensive care unit
length of ICU stay of more than 48 hours | From date of inclusion until 2 days after ICU admission
  duration of ICU stay was greater than 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Flavia R Machado, MD, Principal Investigator — Federal University of São Paulo

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Derived] Machado FR, Cavalcanti AB, Monteiro MB, Sousa JL, Bossa A, Bafi AT, Dal-Pizzol F, Freitas FGR, Lisboa T, Westphal GA, Japiassu AM, Azevedo LCP; Instituto Latino-Americano de Sepsis network investigators. Predictive Accuracy of the Quick Sepsis-related Organ Failure Assessment Score in Brazil. A Prospective Multicenter Study. Am J Respir Crit Care Med. 2020 Apr 1;201(7):789-798. doi: 10.1164/rccm.201905-0917OC. PMID 31910037